CLINICAL TRIAL: NCT04029922
Title: A Phase 1 Open-label, Multicenter Dose Escalation and Expansion Study of MT-5111 in Subjects With Previously Treated Advanced HER2-positive Solid Tumors
Brief Title: Study of MT-5111 in HER2-positive Solid Tumors
Acronym: MT-5111
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study Reprioritization
Sponsor: Molecular Templates, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MT-5111_001
Record Dates: First submitted 2019-07-19; First posted 2019-07-23 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: HER2-positive Solid Cancers

STUDY DESIGN:
Intervention Model Description: MT-5111 (active drug)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A- Dose Escalation (Experimental): Part A- Dose Escalation in patients with previously treated advanced HER2-positive solid tumors.
  The assigned dose level of MT-5111 will be given as an intravenous (IV) infusion over about 30 minutes on the same day every week (i.e., on day 1, day 8 and day 15 of each cycle).
  Interventions: Drug: MT-5111 (experimental study drug)
- Part B- Dose Expansion (Experimental): Part B - Dose Expansion in previously treated HER2-positive breast, GEA and other HER2-positive solid cancers
  Part B will include 3 expansion groups: Group B1 (Breast Cancer) will begin enrolling while Part A is being conducted following the completion of Cohort 7 and Subsequent cohort of subjects in group B1 may enroll into higher doses that are tolerated in Part A. Group B2 (GEA) and Group B3 (Other HER-2 positive solid cancer groups) will begin enrollment after the MTD or RP2D is determined in Part A.
  The assigned dose level of MT-5111 will be given as an intravenous (IV) infusion over about 30 minutes on the same day every week (i.e., on day 1, day 8 and day 15 of each cycle).
  Interventions: Drug: MT-5111 (experimental study drug)

INTERVENTIONS:
Drug: MT-5111 (experimental study drug) — Experimental treatment with MT-5111

SUMMARY:
This will be a Phase 1b, first in human, open-label, dose escalation and expansion study of MT-5111 (a recombinant fusion protein) given as monotherapy in subjects with HER2-positive solid tumors

DETAILED DESCRIPTION:
This study will be conducted in two parts:

Part A (Dose Escalation): The purpose of Part A is to determine the maximum tolerated dose (MTD) or recommended Phase 2 dose (RP2D). Part A will include any type of HER2-positive solid cancer.

Part B (Dose Expansion): The purpose of Part B is to confirm the safety and tolerability of MT-5111 doses selected from those explored in Part A including the MTD or RP2D. Part B will include 3 types of HER2-positive solid cancers in the following 3 expansion groups: Group B1: Breast cancer; Group B2: gastric or gastroesophageal adenocarcinomas (GEA); and Group B3: Other HER2-positive solid cancers.

The Breast Cancer cohort will start enrolling in parallel to Part A.

Up to 178 eligible subjects will be identified and treated through competitive enrollment at multiple study centers globally

In Parts A and B of the study, a subject may participate for the following four periods:

Screening (up to 28 days before first dose of MT-5111)

Treatment period (active period where a subject will receive three weekly doses of MT-5111 over a 21-day treatment cycle)

Short-term Follow-up (30 days after last dose of MT-5111)

Long-term follow-up (up to 24 months after the last dose of MT-5111)

MT-5111 will be given as an intravenous (IV) infusion over about 30 minutes on the same day every week (i.e., on day 1, day 8 and day 15 of each cycle, a cycle being defined as 21 days). A subject can continue receiving MT-5111 as long as it is well-tolerated, their disease has not worsened, or until the subject decides they no longer want to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed, unresectable, locally advanced or metastatic solid cancers:

   * Part A (Dose-Escalation): All HER2-positive solid cancers are eligible
   * Part B (Dose-Expansion): Any type of HER2-positive solid cancer, including breast cancer, and gastric or gastroesophageal adenocarcinomas (GEA).
2. HER2-positive in the latest tumor sample tested for HER2 (testing to be done on a metastatic lesion in cases of metastatic cancers).
3. Relapsed or refractory to or intolerant of existing therapy(ies)
4. At least 1 measurable or evaluable lesion according to RECIST 1.1 (Subjects with evaluable disease only may be included in the dose escalation phase)
5. ECOG performance score of ≤ 1
6. Adequate Bone marrow function as determined by:

   * Absolute neutrophil count (ANC) ≥ 1,000/mm3
   * Platelet count ≥ 75,000 mm³ and
   * Hemoglobin ≥ 8.0 g/dL
   * Red blood cell transfusion within 2 weeks of study treatment start is allowed if hemoglobin levels remain stable
7. Kidney function:

   * Creatinine clearance (CLcr) ≥ 50 mL/min either measured or estimated using the Cockcroft-Gault formula
8. Cardiac Function:

   * Left ventricular ejection fraction (LVEF) ≥ 55% on the echocardiogram (ECHO) assessment (preferred), or multigated acquisition (MUGA) scan, and QTcF ≤ 480 ms for women and QTcF ≤ 450 ms for men [average from three QTcF values on the triplicate 12-lead electrocardiogram (ECG)] at baseline
9. Hepatic function:

   * Total bilirubin ≤ 1.5 x ULN, or ≤ 3 x ULN for subjects with Gilbert's Syndrome and
   * AST ≤ 3 x ULN (or ≤ 5 x ULN if liver metastasis) and ALT ≤ 3 x ULN (or ≤ 5 x ULN if liver metastasis)

Exclusion Criteria:

1. History or current evidence of another tumor that is histologically distinct from the tumor under study
2. Current evidence of new or growing CNS metastases during screening

   * Subjects with known CNS metastases will be eligible if they meet protocol specified criteria
3. Evidence of CTCAE Grade >1 toxicity before the start of treatment, except for hair loss and those Grade 2 toxicities listed as permitted in other eligibility criteria
4. History or evidence of significant cardiovascular disease
5. Current evidence of active, uncontrolled hepatitis B virus, hepatitis C virus, human immunodeficiency virus (HIV) (evidenced by detectable viral load by PCR) or acquired immunodeficiency syndrome (AIDS) related illness
6. Current evidence of ≥ grade 2 underlying pulmonary disease
7. Certain exclusionary prior treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
To evaluate safety and determine the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) | 21 day cycle
  Evaluation of safety of MT-5111 as measured by number of subjects with adverse events using Common Terminology Criteria for Adverse Events (CTCAE) v 5.0
To evaluate tolerability and determine the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) | 21 day cycle
  Evaluation of tolerability of MT-5111 as measured by number of subjects with dose limiting toxicities (DLTs)

SECONDARY OUTCOMES:
PK as measured by concentrations of free MT-5111 (Maximum Plasma Concentration [Cmax]) | Day 1, Day 8, and Day 15 in Each 21-Day cycle
  Evaluation of the pharmacokinetic profile of MT-5111
PK as measured by concentrations of free MT-5111 (Time to reach maximum concentration after drug administration [Tmax]) | Day 1, Day 8, and Day 15 in Each 21-Day cycle
  Evaluation of the pharmacokinetic profile of MT-5111
PK as measured by concentrations of free MT-5111 (Area Under the Curve [AUC]) | Day 1, Day 8, and Day 15 in Each 21-Day cycle
  Evaluation of the pharmacokinetic profile of MT-5111
To evaluate the tumor response to MT-5111 | Screening, approximately every 6 weeks, at End of Treatment and 30 days after the last dose
  Objective response rate (ORR) defined as the proportion of subjects with either a complete response or a partial response as determined by investigator assessment
To evaluate the immunogenicity of MT-5111 | Screening (baseline), Day 1 of each 21 day cycle, at the End of Treatment and the Follow-up Visit
  Immunogenicity as measured by MT-5111 (anti-drug antibody [ADA] titer)
To evaluate the immunogenicity of MT-5111 | Screening (baseline), Day 1 of each 21 day cycle, at the End of Treatment and the Follow-up Visit
  Immunogenicity as measured by MT-5111 (neutralizing antibody [NAb])

OTHER OUTCOMES:
To correlate the pharmacodynamic markers of cancer under study (for breast cancer subjects using historic data, if available) | Screening (baseline)
  The expression of HER2, Estrogen Receptor (ER), Progesterone Receptor (PgR) and Ki67 (exploratory) on the tumor cell analyzed by immunohistochemistry
To correlate the pharmacodynamic markers of cancer under study relationship for MT-5111 using the PK, pharmacodynamics, safety, and tumor response variables. | Screening (baseline), every 6 weeks (± 1 week) and within 7 days of the EoT Visit.
  Serum-HER2 (s-HER2)
If warranted by the study results, to evaluate the exposure-response relationship for MT-5111 | Screening (baseline), every 6 weeks (± 1 week) and within 7 days of the EoT Visit.
  Analyze data collected for all primary, secondary and exploratory endpoints using the PK, pharmacodynamics, safety, and tumor response variables
To evaluate overall Survival | 30 days after last dose, and every 3 months for up to 24 months

CONTACTS AND LOCATIONS:
Locations (30):
- United States (23):
  - Mayo Clinic (Arizona), Phoenix, Arizona
  - St. Joseph Heritage Healthcare, Fullerton, California
  - Cancer and Blood Specialty Clinic, Los Alamitos, California
  - Cedars-Sinai Medical Center, Santa Monica, California
  - UCLA Hematology & Oncology, Santa Monica, California
  - Sarah Cannon Research Institute, Denver, Colorado
  - Sylvester Comprehensive Cancer Center (University of Miami), Coral Gables, Florida
  - South Broward Hospital District d/b/a Memorial Healthcare System, Hollywood, Florida
  - Mayo Clinic (Florida), Jacksonville, Florida
  - Orlando Health, Orlando, Florida
  - South Broward Hospital District d/b/a Memorial Healthcare System, Pembroke Pines, Florida
  - BRCR Medical Center, Plantation, Florida
  - Northwestern University, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic (Minnesota), Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Novant Health Cancer Institute, Charlotte, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Prisma Health, Greenville, South Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Mary Crowley Cancer Research, Dallas, Texas
  - The University of Texas Health Science Center, San Antonio, Texas
- Australia (6):
  - St. Vincent's Hospital Melbourne, Fitzroy, Melbourne, VIC
  - Southern Highlands Cancer Centre, Bowral, New South Wales
  - Macquarie University Hospital (Clinical Trials Unit), Macquarie, New South Wales
  - Cancer Research South Australia, Adelaide, South Australia
  - Sunshine Hospital - Western Health, Saint Albans, Victoria
  - Goulburn Valley Health, Shepparton, Victoria
- New Zealand Clinical Research (Christchurch), Christchurch, New Zealand